CLINICAL TRIAL: NCT02083796
Title: Short-term Effects of Thoracic Manipulation on Scapular Kinematics, Muscle Activity and Pain in Shoulder Impingement. A Randomized Controlled Trial
Brief Title: Short-term Effects of Thoracic Manipulation in Shoulder Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Melina Nevoeiro Haik, Master, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Haik-0607; Ethics Committee 465/2011 (Other Grant/Funding Number: FAPESP / 2013/07120-1)
Record Dates: First submitted 2014-02-04; First posted 2014-03-11 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Shoulder Impingement Syndrome
Keywords: manual therapy; rehabilitation; shoulder; spine
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Shoulder impingement_TSM (Experimental): For the manipulation intervention, the subjects were in a seated position and a thrust technique was performed. If no cavitation was detected with the manipulation, the thrust was repeated up to 3 times.
  Interventions: Procedure: Shoulder impingement_TSM
- Shoulder impingement_sham (Sham Comparator): For the sham intervention, the subjects were positioned in the same seated position with the therapist holding the patient in the same position as for the thrust manipulation. In this position, the therapist applied all the same forces as done for a thrust-manipulation and held that position for a few seconds, but a thrust was not used.
  Interventions: Procedure: Shoulder impingement_sham
- Asymptomatic_TSM (Active Comparator): For the manipulation intervention, the subjects were in a seated position and a thrust technique was performed. If no cavitation was detected with the manipulation, the thrust was repeated up to 3 times
  Interventions: Procedure: Asymptomatic_TSM
- Asymptomatic_sham (Sham Comparator): For the sham intervention, the subjects were positioned in the same seated position with the therapist holding the patient in the same position as for the thrust manipulation. In this position, the therapist applied all the same forces as done for a thrust-manipulation and held that position for a few seconds, but a thrust was not used.
  Interventions: Procedure: Asymptomatic_sham

INTERVENTIONS:
Procedure: Shoulder impingement_TSM — A physiotherapist with 4 years of experience in manual therapy will administer the TSM targeting the middle thoracic spine of the subjects.
  Other Names: Spine manipulation; Spinal manipulation; (Spinal) Thrust
  Arms: Shoulder impingement_TSM
Procedure: Asymptomatic_TSM — A physiotherapist with 4 years of experience in manual therapy administered the TSM targeting the middle thoracic spine of the subjects.
  Other Names: Spine manipulation; Spinal manipulation; (Spinal) Thrust
  Arms: Asymptomatic_TSM
Procedure: Shoulder impingement_sham — A physiotherapist with 4 years of experience in manual therapy administered the sham intervention targeting the middle thoracic spine of the subjects.
  Other Names: Sham spinal manipulation
  Arms: Shoulder impingement_sham
Procedure: Asymptomatic_sham — A physiotherapist with 4 years of experience in manual therapy administered the sham intervention targeting the middle thoracic spine of the subjects.
  Other Names: Sham spinal manipulation
  Arms: Asymptomatic_sham

SUMMARY:
The hypothesis of this study is that thoracic spine manipulation would reduce pain in subjects with SIS and cause changes in scapular kinematics and muscle activity in subjects with impingement symptoms and in asymptomatic subjects. With this study, the investigators want to answer if possible changes in scapular motion and muscle activity following a TSM depend on the symptoms or if it is generic to individuals without shoulder dysfunction and not specific to subjects with shoulder impingement.

DETAILED DESCRIPTION:
Subjects with shoulder impingement signs will be evaluated and will be compared with subjects asymptomatic for shoulder symptoms. Both subjects will be randomly assigned to one of two intervention groups: thoracic spinal manipulation (TSM) or sham intervention. We want to know if possible changes in scapular motion and muscle activity following a TSM depend on the symptoms or if it is generic to everyone. Also, we want to know if TSM reduces shoulder pain immediately and in a short-therm period.

ELIGIBILITY:
Inclusion Criteria (symptomatic subjects): To present with at least 3 of the following findings:

* positive Neer impingement test,
* positive Hawkins impingement test,
* positive Jobe test,
* pain with passive or isometric resisted shoulder lateral rotation,
* pain with active shoulder elevation,
* pain with palpation of rotator cuff tendons,
* pain in the C5 or C6 dermatome region.

Exclusion Criteria (symptomatic subjects):

* signs of "red flags" for spinal manipulation (eg, fracture, osteoporosis, malignancy, infection, and active inflammatory process),
* pregnancy
* systemic illnesses
* if received physical therapy or manual therapy treatment within the 6 months prior to the evaluation
* signs of complete rotator cuff tear or acute inflammation
* cervical-thoracic spine related symptoms (ie, positive cervical compression test and excessive kyphosis)
* scoliosis
* glenohumeral instability (ie, positive apprehension, anterior drawer, or sulcus tests)
* previous upper extremity fracture or shoulder surgery.

Exclusion Criteria (asymptomatic subjects):

* any positive test for shoulder impingement
* signs of "red flags" for spinal manipulation (eg, fracture, osteoporosis, malignancy, infection, and active inflammatory process),
* pregnancy
* systemic illnesses
* if received physical therapy or manual therapy treatment within the 6 months prior to the evaluation
* signs of complete rotator cuff tear or acute inflammation
* cervical-thoracic spine related symptoms (ie, positive cervical compression test and excessive kyphosis)
* scoliosis
* glenohumeral instability (ie, positive apprehension, anterior drawer, or sulcus tests)
* previous upper extremity fracture or shoulder surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in scapular orientation from first to third day | Day 1; day 2; day 3
  3D scapular kinematic (upward/downward rotation; internal/external rotation; anterior/posterior tilt) was assessed pre- and-post thoracic spinal manipulation and sham interventions at first and second days. At the third day of evaluation the measure was assessed only once.

SECONDARY OUTCOMES:
Change in shoulder function from first to third day | Day 1; Day 2; Day 3
  Shoulder function was assessed at the beginning of each data collection day (days 1 to 3) using Disabilities of the Arm, Shoulder and Hand (DASH) and Western Ontario Rotator Cuff Index (WORC) questionnaires.
Change in scapular muscle activity from first to third day | Day 1; Day 2; Day 3
  3D scapular kinematic was assessed pre- and-post thoracic spinal manipulation and sham interventions at first and second days. At the third day of evaluation the measure was assessed only once.
Change in shoulder pain from first to third day | Day 1; Day 2; Day 3
  Shoulder pain was assessed pre- and-post thoracic spinal manipulation and sham interventions at first and second days. At the third day of evaluation the measure was assessed only once.

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Camargo, doctor, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Haik MN, Alburquerque-Sendin F, Camargo PR. Short-Term Effects of Thoracic Spine Manipulation on Shoulder Impingement Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1594-1605. doi: 10.1016/j.apmr.2017.02.003. Epub 2017 Mar 1. PMID 28259517